CLINICAL TRIAL: NCT00553410
Title: SOLE, Study of Letrozole Extension, A Phase III Trial Evaluating the Role of Continuous Letrozole Versus Intermittent Letrozole Following 4 to 6 Years of Prior Adjuvant Endocrine Therapy for Postmenopausal Women With Hormone-Receptor Positive, Node Positive Early Stage Breast Cancer
Brief Title: Letrozole in Preventing Cancer in Postmenopausal Women Who Have Received 4-6 Years of Hormone Therapy for Hormone Receptor-Positive, Lymph Node-Positive, Early-Stage Breast Cancer
Acronym: SOLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IBCSG 35-07 / BIG 1-07; 2007-001370-88 (EudraCT Number); CDR0000574249 (Registry Identifier: CT.gov)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous letrozole (Active Comparator): Continuous letrozole: 5 years continuously (2.5 mg Letrozole daily)
  Interventions: Drug: Letrozole
- Intermittent letrozole (Experimental): Intermittent letrozole: 48 months over 5 yrs: 4 x 9 months (9 mo followed by 3 mo treatment-free interval in yrs 1-4, -> 36 mo) plus 1 x 12 mo in yr 5 -> 48 months
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Film-coated tablet, oral use, 2.5 mg Letrozole daily for 5 years continuously
  Arms: Continuous letrozole
Drug: Letrozole — Film-coated tablet, oral use, 2.5 mg daily, 48 months over 5 yrs: 4 x 9 months (9 mo followed by 3 mo treatment-free interval in yrs 1-4, -> 36 mo) plus 1 x 12 mo in yr 5 -> 48 months
  Arms: Intermittent letrozole

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Letrozole may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known which regimen of letrozole is more effective in postmenopausal women who have received hormone therapy for early-stage breast cancer.

PURPOSE: This randomized phase III trial is comparing two different regimens of letrozole in preventing cancer in postmenopausal women who have received 4-6 years of hormone therapy for hormone receptor-positive, lymph node-positive, early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival (DFS) of postmenopausal women treated with continuous letrozole for 5 years vs intermittent letrozole over a 5-year period.

Secondary

* Compare overall survival of patients treated with these two regimens.
* Compare distant DFS of these patients.
* Compare breast cancer-free interval of these patients.
* Compare sites of first DFS failure in these patients.
* Compare second (nonbreast) malignancies in these patients.
* Compare deaths without prior cancer events in these patients.
* Compare adverse events resulting from these two regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to treatment center and type of prior endocrine therapy (selective estrogen receptor modulators [SERMs] alone vs aromatase inhibitors [AIs] alone vs both SERMs and AIs each for at least 1 month). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral letrozole daily for 5 years.
* Arm II: Patients receive oral letrozole daily for the first 9 months of years 1 through 4, followed by 12 months in year 5.

After completion of study therapy, patients are followed annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of prior operable, noninflammatory breast cancer meeting the following criteria:

  * Steroid hormone receptor-positive tumors (estrogen receptor and/or progesterone receptor), determined by immunohistochemistry, after primary surgery and before commencement of prior endocrine therapy
  * Prior local treatment including surgery with or without radiotherapy for primary breast cancer with no known clinical residual loco-regional disease
  * Following primary surgery, eligible patients must have had evidence of lymph node involvement either in the axillary or internal mammary nodes, but not supraclavicular nodes
  * Clinically disease-free
* Must have completed 4-6 years of prior adjuvant selective estrogen receptor modulators (SERMs), aromatase inhibitors (AIs), or a sequential combination of both

  * When calculating 4-6 years, neoadjuvant endocrine therapy should not be included
* No evidence of recurrent disease or distant metastatic disease
* No prior bilateral breast cancer

PATIENT CHARACTERISTICS:

* Female
* Must be postmenopausal by any of the following criteria:

  * Patients of any age who have had a bilateral oophorectomy (including radiation castration AND amenorrheic for > 3 months)
  * Patients 56 years old or older with any evidence of ovarian function must have biochemical evidence of definite postmenopausal status (defined as estradiol, luteinizing hormone [LH], and follicle-stimulating hormone [FSH] in the postmenopausal range)
  * Patients 55 years old or younger must have biochemical evidence of definite postmenopausal status (defined as estradiol, LH, and FSH in the postmenopausal range)

    * Patients who have received prior luteinizing-hormone releasing-hormone (LHRH) analogues within the last year are eligible if they have definite evidence of postmenopausal status as defined above
* Clinically adequate hepatic function
* No bone fracture due to osteoporosis at any time during the 4-6 years of prior therapy
* No prior or current malignancy except adequately treated basal cell or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, or contra- or ipsilateral in situ breast carcinoma
* No other nonmalignant systemic diseases (cardiovascular, renal, lung, etc.) that would prevent prolonged follow-up
* No psychiatric, addictive, or any other disorder that compromises compliance with protocol requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 12 months since prior and no other concurrent endocrine SERM/AI therapy
* Any type of prior adjuvant therapy allowed including, but not limited to, any of the following:

  * Neoadjuvant chemotherapy
  * Neoadjuvant endocrine therapy
  * Adjuvant chemotherapy
  * Trastuzumab (Herceptin®)
  * Ovarian ablation
  * Gonadotropin releasing hormone analogues
  * Lapatinib ditosylate
* No concurrent hormone-replacement therapy, bisphosphonates (except for treatment of bone loss), or any other investigational agent

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4884 (Actual)
Dates: Start 2007-08; Primary Completion 2018-04 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Colleoni, MD, Study Chair — European Institute of Oncology
Locations (164):
- United States (2):
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
- Australia (17):
  - Armidale Hospital, Armidale, New South Wales
  - Bankstown - Lidcombe Hospital, Bankstown, New South Wales
  - Southern Highlands Cancer Center, Bowral, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Breast Center, Gateshead, New South Wales
  - Port Mcquarie Base Hospital, Port Macquarie, New South Wales
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Tamworth Base Hospital, Tamworth, New South Wales
  - Tweed Heads Hospital, Tweed Heads, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - North West Regional Hospital, Burnie, Tasmania
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Health, Heidelberg, Victoria
  - Maroondah Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (12):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medizinische Universitaet Graz, Graz
  - Innsbruck Universitaetsklinik, Innsbruck
  - Krankenhaus BHS Linz, Linz
  - Allgemeines Krankenhaus Linz, Linz
  - St. Johanns-Spital, Salzburg
  - Medical University of Vienna, Vienna
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
  - Krankenhaus Lainz, Vienna
  - Hanusch-Krankenhaus, Vienna
  - LKH Villach, Villach
  - Klinikum Kreuzschwestern Wels GmbH, Wels
- Belgium (26):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Cliniques du Sud Luxembourg, Arlon
  - Imelda vzw, Ziekenhuis, Bonheiden
  - AZ Klina, Brasschaat
  - Institut Jules Bordet, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Algemeen Ziekenhuis Sint-Maarten - Campus Rooiberg, Duffel
  - Universitair Ziekenhuis Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - Virga Jesse Hospital, Hasselt
  - Centre Hospitalier Hutois, Huy
  - AZ Groeninge - Oncologisch Centrum, Kortrijk
  - U.Z. Gasthuisberg, Leuven
  - Centre Hospitalier de l'Ardenne, Libramont
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Clinique Saint-Joseph, Liège
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Jan Palfijn Hospital, Merksem
  - AZ Damiaan, Ostend
  - Clinique Saint-Pierre, Ottignies
  - Clinique Saint Vincent, Rocourt
  - AZ Nikolaas - Sint-Niklaas, Sint-Niklaas
  - Sint-Elisabethziekenhuis, Turnhout
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- Chile (7):
  - Hospital Santiago Oriente Dr. Luis Tisne Brousse, Peñalolén
  - Fundacion Arturo Lopez Perez, Santiago
  - Hospital Clinico San Borja Arriaran, Santiago
  - Instituto Nacional Del Cancer, Santiago
  - IRAM - Chile, Santiago
  - Hospital Clinico Regional de Valdivia at University Austral de Chile, Valdivia
  - Hospital Carlos Van Buren, Valparaíso
- Denmark (12):
  - Aarhus Universitetshospital - Aarhus Sygehus, Aarhus C
  - Copenhagen County Herlev University Hospital, Copenhagen
  - Centralsygehus Esbjerg, Esbjerg
  - Herning Central Hospital, Herning
  - Hillerod Hospital, Hillerød
  - Naestved Hospital, Næstved
  - Odense University Hospital, Odense
  - Roskilde Amtssygehuset, Roskilde
  - Bornholms Hospital, Rønne
  - Sonderborg Sygehus, Sønderborg
  - Vejle Sygehus, Vejle
  - Viborg Sygehus, Viborg
- Institut Bergonie, Bordeaux, France
- Germany (18):
  - Aalen Breast Center, Aalen
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Allgemeinen Krankenhaus Celle Kinderklinik, Celle
  - Klinikum Deggendorf, Deggendorf
  - Praxis Dr. Wilke - Onkologie am Klinikum Fuerth, Fürth
  - Vinzenzkrankenhaus Hannover gGmbH, Hanover
  - Henriettenstiftung Krankenhaus, Hanover
  - Gynaekologisch-onkologische Praxis Hannover, Hanover
  - Frauenheilkunde u. Geburtshilfe, Ilsede
  - Asklepios Klinik Lich, Lich
  - Gemeinschaftspraxis Gynaekologie & Geburtshilfe, Mannheim
  - Klinikum Meiningen GmbH, Meiningen
  - Klinikum Memmingen, Memmingen
  - Klinikum Offenback GmbH, Offenbach
  - Deaconess Hospital, Schwäbisch Hall
  - Johanniter Kankenhaus Stendal, Stendal
  - SRH Zentralklinikum Suhl GmbH, Suhl
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (2):
  - National Institute of Oncology - Budapest, Budapest
  - Szeged University, Szeged
- Tata Memorial Hospital, Mumbai, India
- Italy (12):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedale degli Infermi - ASL 12, Biella
  - Azienda Sanitaria di Bolzano, Bolzano
  - Spedali Civili di Brescia, Brescia
  - A. Perrino Hospital, Brindisi
  - Azienda Istituti Ospitalieri, Cremona
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - European Institute of Oncology, Milan
  - Fondazione Salvatore Maugeri, Pavia
  - Misericordia e Dolce Hospital, Prato
  - Ospedale Civile Rimini, Rimini
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Japan (7):
  - Osaka Rosai Hospital, Sakai, Osaka
  - Sagara Hospital, Kagoshima
  - Kumamoto University Faculty of Medical and Pharmaceutical Sciences, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Niigata Cancer Center Hospital, Niigata
  - Yao Municipal Hospital, Osaka
  - Tokyo Metropolitan - Komagome Hospital, Tokyo
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Russian Academy of Medical Sciences Cancer Research Center, Moscow, Russia
- South Africa (2):
  - Tygerberg Hospital, Cape Town
  - Sandton Oncology Medical Research, Sandton
- Spain (10):
  - Vall d'Hebron University Hospital, Barcelona
  - M. D. Anderson International Espana SA, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Sant Joan de Reus, Reus
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital de Torrevieja, Torrevieja
  - Instituto Valenciano De Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (6):
  - Lasarettet i Boras, Borås
  - Malarsjukhuset Hospital, Eskilstuna
  - Sahlgrenska University Hospital, Gothenburg
  - Lidkoping Hospital, Lidköping
  - Skaraborgs Hospital, Skövde
  - Karolinska University Hospital - Huddinge, Stockholm
- Switzerland (23):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Oncocare Sonnenhof-Klinik Engeriedspital, Bern
  - AndreasKlinik Cham Zug, Cham
  - Kantonsspital Graubuenden, Chur
  - Brustzentrum Thurgau at Kantonsspital Frauenfeld, Frauenfeld
  - Kantonsspital Freiburg, Fribourg
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Lago Maggiore Oncology Foundation, Locarno
  - Ospedale "la Carita", Locarno, Locarno
  - Ospedale Civico, Lugano
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital Olten, Olten
  - Tumor Zentrum ZeTup St. Gallen und Chur, Sankt Gallen
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopital Regional de Sion-Herens-Conthey, Sion
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - Breast Center, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich
- United Kingdom (2):
  - Borders General Hospital, Melrose, England
  - Dumfries & Galloway Royal Infirmary, Dumfries, Scotland

REFERENCES:
- [Derived] Guerini-Rocco E, Gray KP, Fumagalli C, Reforgiato MR, Leone I, Rafaniello Raviele P, Munzone E, Kammler R, Neven P, Hitre E, Jerusalem G, Simoncini E, Gombos A, Deleu I, Karlsson P, Aebi S, Chirgwin J, Di Lauro V, Thompson A, Graas MP, Barber M, Fontaine C, Loibl S, Gavila J, Kuroi K, Muller B, O'Reilly S, Di Leo A, Goldhirsch A, Viale G, Barberis M, Regan MM, Colleoni M. Genomic Aberrations and Late Recurrence in Postmenopausal Women with Hormone Receptor-positive Early Breast Cancer: Results from the SOLE Trial. Clin Cancer Res. 2021 Jan 15;27(2):504-512. doi: 10.1158/1078-0432.CCR-20-0126. Epub 2020 Oct 20. PMID 33082214
- [Derived] Colleoni M, Luo W, Karlsson P, Chirgwin J, Aebi S, Jerusalem G, Neven P, Hitre E, Graas MP, Simoncini E, Kamby C, Thompson A, Loibl S, Gavila J, Kuroi K, Marth C, Muller B, O'Reilly S, Di Lauro V, Gombos A, Ruhstaller T, Burstein H, Ribi K, Bernhard J, Viale G, Maibach R, Rabaglio-Poretti M, Gelber RD, Coates AS, Di Leo A, Regan MM, Goldhirsch A; SOLE Investigators. Extended adjuvant intermittent letrozole versus continuous letrozole in postmenopausal women with breast cancer (SOLE): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2018 Jan;19(1):127-138. doi: 10.1016/S1470-2045(17)30715-5. Epub 2017 Nov 17. PMID 29158011

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Continuous Letrozole: Continuous letrozole: 5 years continuously (2.5 mg Letrozole daily)
  Letrozole: Film-coated tablet, oral use, 2.5 mg Letrozole daily for 5 years continuously
- Arm B: Intermittent Letrozole: Intermittent letrozole: 48 months over 5 yrs: 4 x 9 months (9 mo followed by 3 mo treatment-free interval in yrs 1-4, -> 36 mo) plus 1 x 12 mo in yr 5 -> 48 months
  Letrozole: Film-coated tablet, oral use, 2.5 mg daily, 48 months over 5 yrs: 4 x 9 months (9 mo followed by 3 mo treatment-free interval in yrs 1-4, -> 36 mo) plus 1 x 12 mo in yr 5 -> 48 months
Period: Overall Study
Arm/Group | Arm A: Continuous Letrozole | Arm B: Intermittent Letrozole
Started | 2441 | 2443
Completed | 2426 | 2425
Not Completed | 15 | 18

BASELINE CHARACTERISTICS:
Population: Randomized patients, regardless of eligibility status; exceptions were patients who immediately withdrew consent prior to treatment initiation and declined all participation, patients determined to be without adequate documentation of informed consent, and/or patients at a participating center determined not to be compliant with protocol procedures
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Continuous Letrozole | Arm B: Intermittent Letrozole | Total
Number analyzed (Participants) | 2426 | 2425 | 4851
Age, Customized [Count of Participants; unit: Participants]
  <55 | 668 | 671 | 1339
  55-59 | 504 | 496 | 1000
  60-64 | 451 | 471 | 922
  65-69 | 400 | 375 | 775
  70+ | 383 | 412 | 795
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2426 | 2425 | 4851
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 2199 | 2211 | 4410
  Black | 10 | 9 | 19
  Asian | 119 | 121 | 240
  Other | 97 | 83 | 180
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Hungary | 78 | 77 | 155
  United States | 21 | 19 | 40
  Japan | 93 | 99 | 192
  United Kingdom | 217 | 216 | 433
  Switzerland | 159 | 159 | 318
  India | 8 | 8 | 16
  Russia | 22 | 21 | 43
  Spain | 137 | 134 | 271
  New Zealand | 10 | 9 | 19
  Austria | 88 | 92 | 180
  Sweden | 104 | 105 | 209
  Belgium | 509 | 520 | 1029
  Denmark | 223 | 218 | 441
  Italy | 287 | 291 | 578
  South Africa | 28 | 28 | 56
  Australia | 182 | 171 | 353
  Chile | 70 | 70 | 140
  France | 14 | 16 | 30
  Peru | 33 | 33 | 66
  Germany | 146 | 145 | 291

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: Duration of time from randomization to the first indication of the following events: invasive recurrence at local (including recurrence restricted to the breast after breast conserving treatment), regional or distant sites; a new invasive cancer in the contralateral breast; any second (non-breast) invasive malignancy; or a death without prior cancer event. Appearance of DCIS or LCIS either in the ipsilateral or in the contralateral breast was not be considered as an event for DFS. In the absence of an event, DFS was censored at the date of last follow-up visit.
Time Frame: 5-year estimates, reported at a median follow-up of 60 months
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A: Continuous Letrozole | Arm B: Intermittent Letrozole
Number analyzed (Participants) | 2426 | 2425
percentage of patients | 87.5 [86 to 88.8] | 85.8 [84.2 to 87.2]
Statistical Analysis 1: Comparison: Arm A: Continuous Letrozole vs Arm B: Intermittent Letrozole; Test type: Superiority; p = .31, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [.93 to 1.26]

2. Secondary Outcome: Overall Survival
Description: Duration of time from randomization to death from any cause, or was censored at the date last known alive. (Note, for patients who withdrew consent or were lost to follow-up but follow-up for survival was possible through hospital or registry records, OS was censored at the date last known alive rather than date of last follow-up/withdrawn consent).
Time Frame: 5-year estimates, reported at a median follow-up of 60 months
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A: Continuous Letrozole | Arm B: Intermittent Letrozole
Number analyzed (Participants) | 2426 | 2425
percentage of patients | 93.7 [92.6 to 94.7] | 94.3 [93.2 to 95.2]
Statistical Analysis 1: Comparison: Arm A: Continuous Letrozole vs Arm B: Intermittent Letrozole; Test type: Superiority; p = .16, Log Rank; Hazard Ratio (HR) = .85, 95% CI 2-sided [.68 to 1.06]

3. Secondary Outcome: Distant Recurrence-free Interval (DRFI)
Description: Duration of time from randomization to the first indication of invasive breast recurrence at a distant site. In the absence of an event, DRFI was censored at the date of last follow-up visit or date or death without distant recurrence.*
  *This endpoint replaced DDFS, which was specified in the protocol
Time Frame: 5-year estimates, reported at a median follow-up of 60 months
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A: Continuous Letrozole | Arm B: Intermittent Letrozole
Number analyzed (Participants) | 2426 | 2425
percentage of patients | 92.5 [91.3 to 93.5] | 93.2 [92 to 94.2]
Statistical Analysis 1: Comparison: Arm A: Continuous Letrozole vs Arm B: Intermittent Letrozole; Test type: Superiority; p = .25, Log Rank; Hazard Ratio (HR) = .88, 95% CI 2-sided [.71 to 1.09]

4. Secondary Outcome: Breast Cancer-free Interval
Description: Duration of time from randomization to the first indication of the following events: invasive breast recurrence at local, regional or distant sites; a new invasive cancer in the contralateral breast (second non-breast malignancies are ignored). In the absence of an event, BCFI was censored at the date of last follow-up visit or date of death without prior breast cancer event.
Time Frame: 5-year estimates, reported at a median follow-up of 60 months
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A: Continuous Letrozole | Arm B: Intermittent Letrozole
Number analyzed (Participants) | 2426 | 2425
percentage of patients | 91.2 [89.9 to 92.3] | 90.9 [89.6 to 92.1]
Statistical Analysis 1: Comparison: Arm A: Continuous Letrozole vs Arm B: Intermittent Letrozole; Test type: Superiority; p = .84, Log Rank; Hazard Ratio (HR) = .98, 95% CI 2-sided [.81 to 1.18]

ADVERSE EVENTS:
Time Frame: during or within 30 days after stopping study treatment
Description: Adverse event is defined as any untoward medical occurrence that occurs from the first dose of study medication until 30 days after final dose, regardless of whether it is considered related to a medication. Any known untoward event that occurs subsequent to the adverse event reporting period that the investigator assesses as possibly related to the protocol treatment should be considered an adverse event. Symptoms of the targeted cancer (if applicable) should not be reported as adverse events.
Arm/Group | Arm A: Continuous Letrozole | Arm B: Intermittent Letrozole
All-Cause Mortality (participants affected / at risk) | 170/2426 | 146/2425
Serious Adverse Events (participants affected / at risk) | 1004/2411 | 1052/2417
Other Adverse Events (participants affected / at risk) | 2257/2411 | 2261/2417
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Continuous Letrozole (N=2411) | Arm B: Intermittent Letrozole (N=2417)
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1
Cardiac Arrhythmia-Other (Specify) (Cardiac disorders) | 2 | 2
Cardiac-ischemia/infarction (Cardiac disorders) | 21 | 22
Conduction abnormality/Atrioventricular heart block - AV block-2nd degree Mobitz Type I (Wenckebach) (Cardiac disorders) | 0 | 2
Conduction abnormality/Atrioventricular heart block - AV block-third degree (complete AV block) (Cardiac disorders) | 2 | 0
Conduction abnormality/Atrioventricular heart block - Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 5 | 3
Pain - Cardiac/heart (Cardiac disorders) | 1 | 0
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 2
Right ventricular dysfunction (cor pulmonale) (Cardiac disorders) | 1 | 2
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 9 | 17
Supraventricular and nodal arrhythmia - Atrial flutter (Cardiac disorders) | 3 | 0
Supraventricular and nodal arrhythmia - Atrial tachycardia/paroxysmal atrial tachycardia (Cardiac disorders) | 2 | 1
Supraventricular and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 0 | 1
Supraventricular and nodal arrhythmia - Supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
Supraventricular and nodal arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Valvular heart disease (Cardiac disorders) | 12 | 6
Ventricular arrhythmia - Ventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 2 | 1
Auditory/Ear-Other (Specify) (Ear and labyrinth disorders) | 3 | 8
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 0 | 1
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 0 | 1
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 | 2
Endocrine-Other (Specify) (Endocrine disorders) | 3 | 2
Cataract (Eye disorders) | 8 | 10
Dry eye syndrome (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 2
Ocular/Visual-Other (Specify) (Eye disorders) | 1 | 3
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 2
Vision-blurred vision (Eye disorders) | 1 | 1
Vision-photophobia (Eye disorders) | 1 | 0
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 0 | 1
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 0 | 1
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 0 | 1
Obstruction, GI - Cecum (Gastrointestinal disorders) | 0 | 1
Obstruction, GI - Esophagus (Gastrointestinal disorders) | 1 | 0
Obstruction, GI - Ileum (Gastrointestinal disorders) | 1 | 0
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1 | 0
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 3 | 2
Dental: teeth (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 5
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 2 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 | 2
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 6 | 4
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 3 | 1
Mucositis/stomatitis (clinical exam) - Anus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 | 3
Pain - Stomach (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 58 | 48
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 | 1
Constitutional Symptoms-Other (Specify) (General disorders) | 0 | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 1 | 2
Death not associated with CTCAE term - Sudden death (General disorders) | 2 | 0
Pain - Chest/thorax NOS (General disorders) | 2 | 1
Pain - Pain NOS (General disorders) | 1 | 0
Pain-Other (Specify) (General disorders) | 1 | 3
Obstruction, GI - Gallbladder (Hepatobiliary disorders) | 1 | 1
Stricture/stenosis (including anastomotic), GI - Biliary tree (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 6 | 13
Hepatobiliary/Pancreas-Other (Specify) (Hepatobiliary disorders) | 5 | 6
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 5 | 1
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Brain (encephalitis, infectious) (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Foreign body (e.g., graft, implant) (Infections and infestations) | 3 | 3
Infection with unknown ANC - Foreign body (e.g., graft, implant, prosthesis, stent) (Infections and infestations) | 0 | 1
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils -Lung (pneumonia) (Infections and infestations) | 1 | 1
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils -Small bowel NOS (Infections and infestations) | 1 | 0
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Kidney (Infections and infestations) | 0 | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Paranasal (Infections and infestations) | 0 | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Pharynx (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Abdomen NOS (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Anal/perianal (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Appendix (Infections and infestations) | 4 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 2 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Bone (osteomyelitis) (Infections and infestations) | 0 | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Brain + Spinal cord (encephalomyelitis) (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Bronchus (Infections and infestations) | 1 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 1 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Colon (Infections and infestations) | 1 | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Gallbladder (cholecystitis) (Infections and infestations) | 2 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Joint (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Kidney (Infections and infestations) | 1 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 6 | 8
Infection with normal ANC or Grade 1 or 2 neutrophils - Lymphatic (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Nerve-peripheral (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 9 | 9
Infection with normal ANC or Grade 1 or 2 neutrophils - Small bowel NOS (Infections and infestations) | 1 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 3 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Wound (Infections and infestations) | 4 | 0
Infection with unknown ANC - Appendix (Infections and infestations) | 0 | 1
Infection with unknown ANC - Dental-tooth (Infections and infestations) | 1 | 0
Infection with unknown ANC - Larynx (Infections and infestations) | 0 | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 7 | 3
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 7 | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 2 | 1
Infection with unknown ANC - Wound (Infections and infestations) | 1 | 1
Infection-Other (Specify) (Infections and infestations) | 1 | 3
Viral hepatitis (Infections and infestations) | 0 | 1
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 66 | 62
Intra-operative injury - Joint (Injury, poisoning and procedural complications) | 0 | 1
Intra-operative injury - Oral (Injury, poisoning and procedural complications) | 1 | 0
Intra-operative injury - Spleen (Injury, poisoning and procedural complications) | 1 | 0
Local complication - device/prosthesis-related (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 18 | 20
Vessel injury-artery - Aorta (Injury, poisoning and procedural complications) | 0 | 1
Vessel injury-artery - Carotid (Injury, poisoning and procedural complications) | 1 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 | 0
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 0 | 1
Coagulation-Other (Specify) (Investigations) | 0 | 1
GGT (gamma-glutamyl transpeptidase) (Investigations) | 1 | 0
INR (International Normalized Ratio of prothrombin time) (Investigations) | 0 | 1
Lipase (Investigations) | 0 | 1
Metabolic/Laboratory-Other (Specify) (Investigations) | 1 | 0
Platelets (Investigations) | 2 | 0
Weight gain (Investigations) | 1 | 2
Weight loss (Investigations) | 1 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 22 | 34
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Obesity (Metabolism and nutrition disorders) | 37 | 42
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 8 | 10
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint-function (Musculoskeletal and connective tissue disorders) | 8 | 12
Lymphedema-related fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 9 | 15
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 17 | 27
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain - Bone (Musculoskeletal and connective tissue disorders) | 58 | 46
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 151 | 139
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 54 | 53
Pain - Neck (Musculoskeletal and connective tissue disorders) | 2 | 0
Soft tissue necrosis - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 | 0
Hemorrhage, CNS (Nervous system disorders) | 7 | 9
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 | 1
Ataxia (incoordination) (Nervous system disorders) | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 31 | 24
Cognitive disturbance (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 10 | 10
Encephalopathy (Nervous system disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 3
Mental status (Nervous system disorders) | 1 | 0
Myelitis (Nervous system disorders) | 1 | 0
Neurology-Other (Specify) (Nervous system disorders) | 12 | 13
Neuropathy: cranial - CN VII Motor-face; Sensory-taste (Nervous system disorders) | 1 | 0
Neuropathy: cranial - CN VIII Hearing and balance (Nervous system disorders) | 1 | 0
Neuropathy: motor (Nervous system disorders) | 1 | 1
Neuropathy: sensory (Nervous system disorders) | 3 | 2
Pain - Head/headache (Nervous system disorders) | 12 | 5
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 2 | 7
Seizure (Nervous system disorders) | 1 | 0
Syncope (fainting) (Nervous system disorders) | 5 | 9
Vasovagal episode (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 59 | 52
Mood alteration - anxiety (Psychiatric disorders) | 2 | 0
Mood alteration - depression (Psychiatric disorders) | 54 | 61
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 | 0
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 | 0
Incontinence, urinary (Renal and urinary disorders) | 2 | 1
Obstruction, GU - Ureter (Renal and urinary disorders) | 0 | 1
Obstruction, GU - Urethra (Renal and urinary disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 5 | 5
Renal/Genitourinary-Other (Specify) (Renal and urinary disorders) | 10 | 12
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 1 | 0
Pain - Pelvis (Reproductive system and breast disorders) | 1 | 0
Sexual/Reproductive Function-Other (Specify) (Reproductive system and breast disorders) | 3 | 4
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstruction/stenosis of airway - Bronchus (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 3 | 3
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 0
Hematoma (Vascular disorders) | 0 | 1
Hemorrhage/Bleeding-Other (Specify) (Vascular disorders) | 0 | 3
Hot flashes/flushes (Vascular disorders) | 70 | 59
Hypertension (Vascular disorders) | 517 | 584
Hypotension (Vascular disorders) | 0 | 1
Peripheral arterial ischemia (Vascular disorders) | 2 | 0
Vascular-Other (Specify) (Vascular disorders) | 3 | 3
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Continuous Letrozole (N=2411) | Arm B: Intermittent Letrozole (N=2417)
Cardiac-ischemia/infarction (Cardiac disorders) | 15 | 23
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1025 | 954
Fracture (Injury, poisoning and procedural complications) | 148 | 136
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 8 | 9
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1113 | 1119
Pain - Bone (Musculoskeletal and connective tissue disorders) | 634 | 613
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1506 | 1453
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 841 | 818
Hemorrhage, CNS (Nervous system disorders) | 4 | 4
CNS cerebrovascular ischemia (Nervous system disorders) | 11 | 8
Insomnia (Psychiatric disorders) | 983 | 961
Mood alteration - depression (Psychiatric disorders) | 767 | 762
Hot flashes/flushes (Vascular disorders) | 1240 | 1217
Hypertension (Vascular disorders) | 539 | 493

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2007-06-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT00553410/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT00553410/SAP_001.pdf